CLINICAL TRIAL: NCT02493491
Title: Neurogenic Dysphonia/Dysphagia Registry
Acronym: StrongVoice
Status: Terminated | Type: Observational
Sponsor: Merz North America, Inc. (Industry)
Collaborators: Carelon Research (Other); Cmed Clinical Services (Other)
Responsible Party: Sponsor
Other Study IDs: METIS M930901001; WI P150999
Record Dates: First submitted 2015-06-30; First posted 2015-07-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Neurogenic Dysphonia; Neurogenic Dysphagia
Keywords: dysphonia; dysphagia; neurogenic; vocal fold augmentation; VFA; vocal fold insufficiency; Prolaryn; Radiesse; Coaptite; voice; Parkinson's Disease; Multiple Sclerosis; Amyotrophic Lateral Sclerosis; ALS; MS; calcium hydroxylapatite; hyaluronic acid
MeSH Terms: conditions — Dysphonia; Deglutition Disorders; Parkinson Disease; Multiple Sclerosis; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Neurogenic Dysphonia/Dysphagia Registry is designed to be purely observational (i.e. non-interventional, exploratory). Patient data collected from the registry is expected to be consistent with any information which can be obtained during usual care of patients with dysphonia/dysphagia treated with vocal fold augmentation.

DETAILED DESCRIPTION:
The Neurogenic Dysphonia/Dysphagia Registry is a 510K post-clearance multicenter, observational, open-label registry of the benefits and risks of management and outcomes of patients with neurogenic dysphonia/dysphagia who have received vocal fold augmentation (VFA).

Enrollment is open to all eligible patients meeting all of the inclusion and none of the exclusion criteria, with a target of 400 patients. Up to 100 sites in the US and abroad will be a part of the registry. Sites will provide retrospective data for active patients who have undergone VFA within the past 24 months at the site and also begin to prospectively enroll patients who are receiving VFA as a part of their usual care. Patients will be followed for up to five years prospectively, until lost to follow-up, or death.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, ≥18 years of age
* Diagnosis of neurogenic dysphonia/dysphagia
* Under active treatment with VFA and follow-up care

Exclusion Criteria:

• Patients with:

* Vocal fold scar
* Laryngeal cancer defect
* Irradiation to the larynx
* Laryngeal trauma
* End-stage cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with neurogenic dysphonia/dysphagia treated with vocal fold augmentation
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Collect and characterize the different types (and frequency) of initial assessments/evaluations performed on patients. | 1 day
  Characterize the initial assessment (e.g. types of assessments/evaluations performed and severity of voice, swallowing, cough as determined by patient reported outcomes where available)
Collect and characterize the different types (and frequency) of subsequent management of neurogenic dysphonia/dysphagia patients who receive VFA in terms of product used, evaluations performed and referrals and recommendations for further treatment | 5 years
  Characterize subsequent management of neurogenic dysphonia/dysphagia patients who receive VFA in terms of product used, evaluations performed and referrals and recommendations for further treatment

SECONDARY OUTCOMES:
Collect patient reported outcomes (PRO) and clinician assessments to characterize voice, swallowing, and cough outcomes post-injection | 5 years
  Characterize voice, swallowing, and cough outcomes post-injection, as determined by patient reported outcomes (PRO) and clinician assessment, as well as select adverse events/complications of interest, associated with use of VFA products in patients with neurogenic dysphonia/dysphagia, including in patients with multiple injections
Collect types and frequency of different patient characteristics and medical care practices associated with improved health outcomes after VFA | 5 years
  Identify patient characteristics and medical care practices associated with improved health outcomes after VFA
Collect and measure information on the duration of effect of Prolaryn products and the need for re-injection | 5 years
  Assess and measure the duration of effect of Prolaryn products
Collect characteristics, management, and outcomes of patients who receive CaHA implants and thryoplasty | 5 years
  Describe characteristics, management, and outcomes of patients who receive CaHA implants and thyroplasty

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sykes, MD, Study Director — Merz North America, Inc.
Locations (12):
- United States (12):
  - Merz Clinical Site, La Jolla, California
  - Merz Clinical Site, Sacramento, California
  - Merz Clinical Site, Augusta, Georgia
  - Merz Clinical Site, Boston, Massachusetts
  - Merz Clinical Site, Burlington, Massachusetts
  - Merz Clinical Site 0010334, New York, New York
  - Merz Clinical Site 0010068, New York, New York
  - Merz Clinical Site 0010333, Sleepy Hollow, New York
  - Merz Clinical Site, Durham, North Carolina
  - Merz Clinical Site 0010332, Pittsburgh, Pennsylvania
  - Merz Clinical Site, Houston, Texas
  - Merz Clinical Site, Norfolk, Virginia